CLINICAL TRIAL: NCT04704713
Title: A Phase III, Randomised, Double Blind, Placebo Controlled, Parallel Group Study, to Evaluate the Safety and Efficacy of Subcutaneous Implants of Afamelanotide (16 mg) in Patients Suffering From Polymorphic Light Eruption (PLE)
Brief Title: Afamelanotide in Patients Suffering From Polymorphic Light Eruption (PLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUV032
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Polymorphic Light Eruption
MeSH Terms: interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Afamelanotide (Experimental): Afamelanotide implants were administered on Days 0 and 60. Patients returned to the clinic on Day 120 for the final visit.
  Interventions: Drug: Afamelanotide
- Placebo (Placebo Comparator): Placebo implants were administered on Days 0 and 60. Patients returned to the clinic on Day 120 for the final visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide
  Arms: Afamelanotide
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study was to evaluate the safety and efficacy of afamelanotide in patients suffering from polymorphic light eruption (PLE).

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than 18 years
* Male or female patients with a documented history of PLE diagnosed or confirmed by a photodermatologist or photobiologist, with a history of PLE related pruritus symptoms.
* Recurrent PLE episodes that occur at least once a year (as evidenced by PLE related pruritus symptoms) developing in their own country (to exclude patients affected only when traveling to sunnier climates)
* Written informed consent prior to the performance of any study-specific procedure
* Are willing and able to comply with the conditions specified in the protocol and study procedures in the opinion of the Investigator

Exclusion Criteria:

* Currently requiring treatment with systemic immunosuppressive agents
* Documented history of other photosensitivity conditions which may be confused with PLE or interfere with the assessment of PLE episodes
* Solarium use in the three months prior to study involvement and throughout the duration of the study
* Use of immunosuppressive medications, drugs that cause hyperpigmentation or any other treatment that in the opinion of the Investigator may interfere with this study
* Documented presence (> 1 in 320) of Anti-Nuclear Antibody (ANA) and/or positive Extractable Nuclear Antibody (ENA); historical results from the 3 years prior to randomisation are acceptable if available
* In the opinion of the Investigator, any evidence of clinically significant organ dysfunction, or any clinically significant deviation from normal in clinical or laboratory parameters
* History of drug or alcohol abuse (in the last 1 year)
* Female who is pregnant (confirmed by positive serum beta-Human chorionic gonadotropin (β-HCG) pregnancy test prior to baseline) or lactating
* Female of child-bearing potential (pre-menopausal, not surgically sterile) that is not using or is not willing to use adequate contraceptive measures (e.g. oral contraceptives, condoms, diaphragm plus spermicide, intrauterine device)
* Sexually active men with partners of child bearing potential not willing to use barrier contraception during the trial and for a period of three months thereafter
* Participation in a clinical trial with another Investigational Medicinal Product (IMP) within 30 days prior to the Screening visit or during the study
* Hypersensitivity to afamelanotide or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05-05 (Actual); Primary Completion 2010-12-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Afamelanotide: Afamelanotide implants were administered on Days 0 and 60. Patients returned to the clinic on Day 120 for the final visit.
  Afamelanotide
- Placebo: Placebo implants were administered on Days 0 and 60. Patients returned to the clinic on Day 120 for the final visit.
  Placebo
Period: Overall Study
Arm/Group | Afamelanotide | Placebo
Started | 15 | 16
Completed | 11 | 12
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afamelanotide | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Severity of PLE Related Pruritus Recorded Using an 11-point Likert Scale
Description: PLE related pruritus was recorded in paper patient diaries commencing using an 11-point Likert scale from 0 (no pruritus) to 10 (most severe pruritus).
Time Frame: From Day 0 to Day 120
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 15 | 16
score on a scale | 0.25 [0.0 to 1.4] | 0.47 [0.0 to 4.1]

2. Secondary Outcome: Frequency (Number) of Documented PLE Episodes Recorded in Paper Patient Diaries
Time Frame: From Day 0 to Day 120
Reporting Status: Not Posted

3. Secondary Outcome: Duration of PLE Episodes Recorded in Paper Patient Diaries
Time Frame: From Day 0 to Day 120
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life Using the Dermatology Life Quality Index (DLQI)
Description: The DLQI questionnaire consists of 10 questions, each answered on a categorical scale. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: At Day 0, Day 60 and Day 120
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Afamelanotide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 7/15 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=15) | Placebo (N=16)
dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Device expulsion (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Influenza (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No